CLINICAL TRIAL: NCT03187743
Title: Personalised Pharmacological Approach to the Tapering of Corticosteroid Doses in Systemic Lupus Patients Treated With Prednisone
Acronym: DECOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160935J; 2017-002050-36 (EudraCT Number)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus erythematosus; Systemic; Corticosteroid; Prednisone; Pharmacokinetics
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetics/dynamics (Experimental): Blood samples at 3 visits
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples at 3 visits :
  V0 : - 5 mL in heparin tube / Pharmacokinetics + Gene Expression Analysis
  V1 : - 5 mL in heparin tube / sample (2 to 5 samples) Pharmacokinetics + Pharmacogenetics + Gene Expression Analysis
  V2 : - 5 mL in heparin tube / Pharmacokinetics + Gene Expression Analysis and - 5 mL in EDTA tube / DNA bank

SUMMARY:
This research study is a multicentre prospective pharmacokinetic study. The clinical and biological data will be collected in the framework of a prospective study. The drug to be evaluated is a glucocorticoid routinely used to treat Systemic lupus erythematosus (SLE) patient. Initial dose of prednisone must be oral and at least 0.5mg/Kg/day, but the precise dosage and the tapering regimen will be determined according to the clinical judgment of the investigator. The duration of the research period for each patient will be 3 months. Three visits (which are all usual care visits) will be needed within the 3 months of the study for collecting data and/or blood sampling

DETAILED DESCRIPTION:
Until now, glucocorticoids always play a leading role in the lupus treatment, and the lupus's prognosis has been greatly improved by the treatment of serious flare-ups with a combination of high-dose corticosteroids and immunosuppressants, notably mycophenolate mofetil (MMF) together with hydroxychloroquine (Plaquenil), survival at 10 years being 70 to 90%. However, corticosteroid treatment is also a major cause of morbidity and mortality, and with 60 years of experience, consensus about "appropriate" dosages, route of administration and tapering regimes has not been reached. In addition, there is a large variability in clinical response to corticosteroid therapy which may be attributed to heterogeneity of SLE, drugs interaction or to environmental and genetic factors, especially to polymorphism of the MDR (multi-drug resistance) -1 and NR3C1 (glucocorticoid nuclear receptor subfamily 3, group C, member 1). There are no previous studies investigating the role of MDR-1 and NR3C1 genes polymorphisms in the response to corticosteroids in lupus patients Drug monitoring of immunosuppressive drugs has been largely explored in renal transplantation and in a lesser extend in SLE (especially for mycophenolic acid). Relationship between prednisolone PK and clinical efficacy/toxicity have been also shown previously especially in renal transplant population. In patients with SLE, only two small series (8 children, 25 adults) have explored this relationship, and suggested that SLE activity and corticosteroid toxicity might be related to prednisolone AUC. Thus, limited data suggest that prednisone monitoring may optimize treatment efficacy and minimize adverse events.

The DECOR study will aim :

1. to search for relationship between prednisolone PK and SLE disease activity in a large series of patients in order to improve the rational of prednisone doses in lupus patients
2. to identify pharmacogenetic factors influencing the response to steroid in order to identify patients sharing a high probability of being responders or resistant to corticosteroids.

This approach could be applied to all inflammatory diseases requiring prolonged corticosteroid treatment, and thus, be a major progress in the use of this old treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 6 years
* Patient who met the American College of Rheumatology criteria (ACR) or the Systemic Lupus International Collaborating Clinics Classification (SLICC) for systemic lupus erythematosus.
* Patients needs (re)initiation of oral prednisone regimen at least at 0.5 mg/Kg/d(or >30mg/d for patients >60 kg) in combination with mycophenolate mofetyl or mycofenolic acid or cyclophosphamide at usual dose including :

  i) patient who receives bolus of methylprednisolone the week before and/or the week after inclusion for treating the lupus flare ii) patient who was previously treated by a low-prednisone dose (≤ 7.5 mg/d in patients ≥ 60 kg and ≤ 0.1 mg/kd/d in patient < 60 kg).

iii) patient who was previously treated by prednisone ≥ 0,5 mg/kg/d (or >30mg/d for patients >60 kg) but stopped since at least one month before inclusion

* Patient with stable doses of other immunosuppressive or biological drugs before inclusion (at least 15 days for Imurel, Methotrexate, Tacrolimus ; at least 6 months for Rituximab, Belimumab) and during the 3 months of patient participation in the study.
* Signed informed consent form by the patient (if aged ≥ 18 years), or by the parents / legal guardian and patient's agreement (if aged < 18 years)
* Patient affiliated to the health insurance system

Exclusion Criteria:

* Patient presents contraindications to corticosteroids
* Patient presents contraindications to MMF, mycofenolic acid or cyclophosphamide for patient receiving immunosupressor
* Patient cannot be treated by oral way
* Patient whose physician has planned to stop prednisone in less than 3 months
* Patient (or parents for minor) are unable to give a written informed consent for physical or psychical reasons
* Patient disagrees with the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
SELENA-SLEDAI score | 3 months

SECONDARY OUTCOMES:
Primary parameters : volume of distribution | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Primary parameters : elimination clearance | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Primary parameters : absorption constant | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Secondary parameters : trough concentration | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Secondary parameters : maximum concentration | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Secondary parameters : Area Under Curve (AUC) | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Secondary parameters : elimination half-life | Day 0, 1 month, 3 months
  To study the pharmacokinetics of prednisolone in a population of patients with SLE
Occurrence of adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michaela SEMERARO, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czock D, Keller F, Rasche FM, Haussler U. Pharmacokinetics and pharmacodynamics of systemically administered glucocorticoids. Clin Pharmacokinet. 2005;44(1):61-98. doi: 10.2165/00003088-200544010-00003. PMID 15634032
- [Background] Sagcal-Gironella AC, Sherwin CM, Tirona RG, Rieder MJ, Brunner HI, Vinks AA. Pharmacokinetics of prednisolone at steady state in young patients with systemic lupus erythematosus on prednisone therapy: an open-label, single-dose study. Clin Ther. 2011 Oct;33(10):1524-36. doi: 10.1016/j.clinthera.2011.09.015. Epub 2011 Oct 7. PMID 21982386
- [Background] Piotrowski P, Burzynski M, Lianeri M, Mostowska M, Wudarski M, Chwalinska-Sadowska H, Jagodzinski PP. Glucocorticoid receptor beta splice variant expression in patients with high and low activity of systemic lupus erythematosus. Folia Histochem Cytobiol. 2007;45(4):339-42. PMID 18165172
- [Background] Du J, Li M, Zhang D, Zhu X, Zhang W, Gu W, Feng Y, Zhai X, Ling C. Flow cytometry analysis of glucocorticoid receptor expression and binding in steroid-sensitive and steroid-resistant patients with systemic lupus erythematosus. Arthritis Res Ther. 2009;11(4):R108. doi: 10.1186/ar2763. Epub 2009 Jul 14. PMID 19594946
- [Background] Stahn C, Lowenberg M, Hommes DW, Buttgereit F. Molecular mechanisms of glucocorticoid action and selective glucocorticoid receptor agonists. Mol Cell Endocrinol. 2007 Sep 15;275(1-2):71-8. doi: 10.1016/j.mce.2007.05.019. Epub 2007 Jun 2. PMID 17630118
- [Background] Derijk RH, de Kloet ER. Corticosteroid receptor polymorphisms: determinants of vulnerability and resilience. Eur J Pharmacol. 2008 Apr 7;583(2-3):303-11. doi: 10.1016/j.ejphar.2007.11.072. Epub 2008 Jan 30. PMID 18321483
- [Background] Mwinyi J, Wenger C, Eloranta JJ, Kullak-Ublick GA. Glucocorticoid receptor gene haplotype structure and steroid therapy outcome in IBD patients. World J Gastroenterol. 2010 Aug 21;16(31):3888-96. doi: 10.3748/wjg.v16.i31.3888. PMID 20712049
- [Background] Nicolaides NC, Galata Z, Kino T, Chrousos GP, Charmandari E. The human glucocorticoid receptor: molecular basis of biologic function. Steroids. 2010 Jan;75(1):1-12. doi: 10.1016/j.steroids.2009.09.002. Epub 2009 Oct 7. PMID 19818358
- [Background] van Rossum EFC, van den Akker ELT. Glucocorticoid resistance. Endocr Dev. 2011;20:127-136. doi: 10.1159/000321234. Epub 2010 Dec 16. PMID 21164266
- [Background] Duru N, van der Goes MC, Jacobs JW, Andrews T, Boers M, Buttgereit F, Caeyers N, Cutolo M, Halliday S, Da Silva JA, Kirwan JR, Ray D, Rovensky J, Severijns G, Westhovens R, Bijlsma JW. EULAR evidence-based and consensus-based recommendations on the management of medium to high-dose glucocorticoid therapy in rheumatic diseases. Ann Rheum Dis. 2013 Dec;72(12):1905-13. doi: 10.1136/annrheumdis-2013-203249. Epub 2013 Jul 19. PMID 23873876
- [Background] Luijten RK, Fritsch-Stork RD, Bijlsma JW, Derksen RH. The use of glucocorticoids in systemic lupus erythematosus. After 60 years still more an art than science. Autoimmun Rev. 2013 Mar;12(5):617-28. doi: 10.1016/j.autrev.2012.12.001. Epub 2012 Dec 8. PMID 23232124
- [Background] Fangtham M, Petri M. 2013 update: Hopkins lupus cohort. Curr Rheumatol Rep. 2013 Sep;15(9):360. doi: 10.1007/s11926-013-0360-0. PMID 23888367
- [Background] Zonana-Nacach A, Barr SG, Magder LS, Petri M. Damage in systemic lupus erythematosus and its association with corticosteroids. Arthritis Rheum. 2000 Aug;43(8):1801-8. doi: 10.1002/1529-0131(200008)43:83.0.CO;2-O. PMID 10943870
- [Background] Al Sawah S, Zhang X, Zhu B, Magder LS, Foster SA, Iikuni N, Petri M. Effect of corticosteroid use by dose on the risk of developing organ damage over time in systemic lupus erythematosus-the Hopkins Lupus Cohort. Lupus Sci Med. 2015 Mar 11;2(1):e000066. doi: 10.1136/lupus-2014-000066. eCollection 2015. PMID 25861455